CLINICAL TRIAL: NCT01445600
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance (PMS) to Monitor the Safety and Efficacy of ALTARGO(Retapamulin) Administered in Korean Patients According to the Prescribing Information
Brief Title: ALTARGO(Retapamulin) PMS(Post-marketing Surveillance)
Acronym: ALTARGOPMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115579
Record Dates: First submitted 2011-09-21; First posted 2011-10-04 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Skin Infections, Bacterial
Keywords: Impetigo; secondarily-infected traumatic lesions; retapamulin
MeSH Terms: conditions — Cellulitis; Impetigo | interventions — retapamulin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALTARGO(retapamulin): The subjects with bacterial skin and skin structure infections (SSSI)
  Interventions: Drug: ALTARGO(retapamulin)

INTERVENTIONS:
Drug: ALTARGO(retapamulin) — Basically there is no treatment allocation. Subjects who would be administered of ALTARGO(retapamulin) at their physicians' discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
This is an open label, multi-centre, non-interventional post-marketing surveillance.

DETAILED DESCRIPTION:
This is an open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety of ALTARGO(retapamulin) treated in Korean patients according to the prescribing information.

ALTARGO is a trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must satisfy the following criteria at study entry:

  1. Subjects administered with ALTARGO(retapamulin) in the topical treatment of the following bacterial skin and skin structure infections (SSSI)
  2. Subjects who the investigator believes that they can and will comply with the requirements of the protocol and follow the administration regimen
  3. Subjects administered with ALTARGO(retapamulin) following the locally approved prescribing information

Exclusion Criteria:

* Considering the nature of observational study, GSK Korea encourages the doctors participating in this study to enrol the subjects prescribed with retapamulin following the locally approved Prescribing Information.

  1. Subjects with a known or suspected hypersensitivity to ALTARGO(retapamulin) or any component of the ointment
  2. Infants under nine months of age

Min Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated ALTARGO(retapamulin) with primary impetigo or secondarily infected traumatic lesions in Korea
Sampling Method: Probability Sample
Enrollment: 3612 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The number of adverse event after ALTARGO(retapamulin) treatment | 14 days

SECONDARY OUTCOMES:
The number of unexpected adverse event after ALTARGO(retapamulin) treatment | 14 days
The number of serious adverse event after ALTARGO(retapamulin) treatment | 14 days
Effectiveness of ALTARGO(retapamulin) treatment | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea